CLINICAL TRIAL: NCT04222946
Title: Stabilometry and Plantar Pressures Changes After Bilateral Dry Needling in Flexor Digitoum Brevis.A Pretest Posttest Study.
Brief Title: Stabilometry and Plantar Pressures Changes After Dry Needling in Flexor Digitoum Brevis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2706201911419
Record Dates: First submitted 2020-01-05; First posted 2020-01-10 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Foot; Dry Needling
Keywords: Stabilometry; Platform; Dry needling; trigger point
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Pretest posttest of bilateral Flexor digitorum Brevis dry neddling intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: (Experimental): bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle

SUMMARY:
The aim of this clinical trial is to check the effects of dry needling in the Flexor digitorum Brevis .

DETAILED DESCRIPTION:
Fiveteen healthy subjects wil be recruited for a quasi-experimental study. Participants will be from 18 to 40 years old, not obese. Participants will be measured before and after bilateral dry neddling in Flexor digitorum Brevis. The investigators will measure stabilometry variables and static footprint. The footprint variables will be divided in bilateral rear foot, bilateral midfoot, bilateral fore foot.

Measures. Stabilometry will be measured by displacement of the center of pressures in X and Y with eyes open and closed , center of pressure (COP) with eyes open and closed, COP area with eyes open and closed, COP antero-posterior (a-p) and medio-lateral (m-lat) directions with eyes open and closed, and COP speed. Two trials will be recorded for each condition and the order of the conditions will be randomized across subjects, eyes open and eyes closed. Foot plantar pressure and surface area of two static footprints will be measured during bipedal standing. Static plantar pressure will be evaluated by means of maximum pressure, medium pressure and surface area of each aspect of the foot (rearfoot, midfoot, and fore foot).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Must have latent trigger point in Flexor Brevis Digitorum muscles

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm
* Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Static footprint | Through study completion, an average of 1 month
  Static footprint will measure plantar presures and surface area of rear food, midfoot and fore foot. Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes open.
Stabilometry variables eyes open | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X and Y with open eyes, Center of Pressure (COP) area and anteroposterior(a-p) and mediolateral directions: COP speed.
Stabilometry variables eyes closed | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X and Y with closed eyes, Center of Pressure (COP) area and anteroposterior(a-p) and mediolateral directions: COP speed.

SECONDARY OUTCOMES:
Static footprint after intervention | Through study completion, an average of 1 month
  Static footprint will measure plantar presures and surface area of rear food, midfoot and fore foot. Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes open.
Stabilometry variables eyes open after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X and Y with open eyes, Center of Pressure (COP) area and anteroposterior(a-p) and mediolateral directions: COP speed.
Stabilometry variables eyes closed after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X and Y with closed eyes, Center of Pressure (COP) area and anteroposterior(a-p) and mediolateral directions: COP speed.

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jimenez, Principal Investigator — Mayuben Clinic
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvioli S, Guidi M, Marcotulli G. The effectiveness of conservative, non-pharmacological treatment, of plantar heel pain: A systematic review with meta-analysis. Foot (Edinb). 2017 Dec;33:57-67. doi: 10.1016/j.foot.2017.05.004. Epub 2017 Jun 15. PMID 29126045
- [Background] David JA, Sankarapandian V, Christopher PR, Chatterjee A, Macaden AS. Injected corticosteroids for treating plantar heel pain in adults. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009348. doi: 10.1002/14651858.CD009348.pub2. PMID 28602048
- [Background] Salom-Moreno J, Sanchez-Mila Z, Ortega-Santiago R, Palacios-Cena M, Truyol-Dominguez S, Fernandez-de-las-Penas C. Changes in spasticity, widespread pressure pain sensitivity, and baropodometry after the application of dry needling in patients who have had a stroke: a randomized controlled trial. J Manipulative Physiol Ther. 2014 Oct;37(8):569-79. doi: 10.1016/j.jmpt.2014.06.003. Epub 2014 Sep 8. PMID 25199825
- [Background] Cotchett MP, Munteanu SE, Landorf KB. Effectiveness of trigger point dry needling for plantar heel pain: a randomized controlled trial. Phys Ther. 2014 Aug;94(8):1083-94. doi: 10.2522/ptj.20130255. Epub 2014 Apr 3. PMID 24700136
- [Background] McNally EG, Shetty S. Plantar fascia: imaging diagnosis and guided treatment. Semin Musculoskelet Radiol. 2010 Sep;14(3):334-43. doi: 10.1055/s-0030-1254522. Epub 2010 Jun 10. PMID 20539958